CLINICAL TRIAL: NCT00923481
Title: A Broad Multi-Histology Phase II Study of the Multi-Kinase Inhibitor R935788 (Fostamatinib Disodium) in Advanced Colorectal, Non-Small Cell Lung, Head and Neck, Hepatocellular and Renal Cell Carcinomas and Pheochromocytoma and Thyroid Tumors
Brief Title: A Broad Multi-histology Phase II Study of the Multi-Kinase Inhibitor R935788 (Fostamatinib Disodium) in Advanced Colorectal, Non-small Cell Lung, Head and Neck Hepatocellular and Renal Cell Carcinomas, and Pheochromocytoma and Thyroid Tumors (Multi-H...
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Shivaani Kummar, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090138; 09-C-0138; NCT00907647 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Neoplasms; Pheochromocytoma; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell
Keywords: Multi-Kinase Inhibitor; Neoplasms; Advanced Cancer; Kidney Cancer; Liver Cancer; Pheochromocytoma; Non-Small Cell Lung Cancer; Colorectal Cancer; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pheochromocytoma; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Neoplasms; Kidney Neoplasms; Liver Neoplasms | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multi-kinase inhibitor Fostamatinib Disodium (R935788) (Experimental): 200 mg BID was the administered dose for the initial part of the study and then a phase I dose escalation was added with 100 mg as the starting dose.
  Interventions: Drug: Fostamatinib disodium

INTERVENTIONS:
Drug: Fostamatinib disodium — 200 mg BID was the administered dose for the initial part of the study and then a phase I dose escalation was added with 100 mg as the starting dose.
  Other Names: R9355788

SUMMARY:
Background:

* The drug R935788 (fostamatanib disodium) is a kinase inhibitor (i.e., it interferes with cell communication and growth and may prevent tumor growth).
* R935788 has shown promising activity in NCI-60 (a panel of 60 diverse human cancer cell lines) against colon cancer, non-small cell lung cancer, and renal cell carcinoma cell lines, as well as in two renal cell xenograft models.
* This is an open-label, Phase II study of R935788. Phase I studies in patients with immune thrombocytopenic purpura, rheumatoid arthritis, and lymphoma have demonstrated safety with a continuous dosing schedule, and a maximum tolerated dose has been established.

Objectives:

* To test an experimental drug called R935788 (fostamatinib disodium) for its ability to stop cancer growth signals, thus slowing the growth of cancer cells in laboratory testing.
* To determine the clinical response of R935788 administered orally twice a day on a continuous schedule in patients with colorectal carcinoma, pheochromocytoma, follicular or papillary thyroid cancer, non-small cell lung cancer, hepatocellular, carcinoma of the head and neck, and renal cell carcinoma.
* To evaluate the effects, safety, and biochemical response of R935788 therapy.

Eligibility:

* Patients with colorectal carcinoma, pheochromocytoma, follicular or papillary thyroid cancer, non-small cell lung cancer (excluding squamous cell histology), hepatocellular cancer, carcinoma of the head and neck, and renal cell carcinoma whose disease has progressed after any therapy or who have no acceptable standard treatment options.
* Patients must have recovered from toxicities of prior therapies to at least eligibility levels.
* Patients who have received radiation or chemotherapy within 4 weeks of study enrollment are not eligible.
* Women who are pregnant or breastfeeding are not eligible.

Design:

* Researchers will conduct the following tests and procedures during the study:

  * Clinic visits with a physical exam, including vital signs and blood pressure, every other week during cycle 1, and once a month starting with cycle 2.
  * Blood will be drawn weekly during cycle 1, every other week during cycle 2, and once a month starting with cycle 3; urine tests will be conducted depending on results of blood tests.
  * Imaging tests, such as computed tomography (CT) scans (a series of x-rays) or ultrasound (an examination using sound waves), will be done every 8 weeks while the patient is receiving R935788.
* R935788 will be administered orally twice a day for 28 days (one cycle). Imaging studies will be obtained every two cycles. Patients will fill in a diary to show when they took the medication and to note any side effects. The 28-day treatment cycle will be repeated as long as the patient is tolerating R935788 and the cancer is either stable or getting better.
* Researchers will conduct the following additional tests to see how the study is affecting the patient:

  * Other research blood samples will be collected before treatment, at cycle 1 week 3, at the beginning of cycle 2, and at 8 weeks.
  * Optional tumor biopsies will be requested before starting treatment, at cycle 1 day 28.
  * Patients with specific lesions or tumors may be asked for an optional tumor biopsy on day 8.

DETAILED DESCRIPTION:
BACKGROUND

* R935788 (fostamatanib disodium) is a kinase inhibitor with activity in vitro against several kinases known to be mutated or aberrantly expressed in malignant cells.
* Anticancer drugs that target multiple kinases are of particular interest because tumors may rely on several different kinase pathways for survival.
* R935788 has shown promising activity in the NCI 60-cell line panel against colon cancer, non-small cell lung cancer, and renal cell carcinoma cell lines, as well as in two renal cell xenograft models. R935788 is orally absorbed in tumor-bearing mice at concentrations that achieve antitumor activity and are not associated with observable toxicity.
* Phase I studies in patients with immune thrombocytopenic purpura, rheumatoid arthritis and lymphoma have demonstrated safety with a continuous dosing schedule, and a maximum tolerated dose (MTD) has been established.

OBJECTIVES

* To determine the clinical response of R935788 administered orally twice a day on a continuous schedule in patients with colorectal carcinoma, pheochromocytoma, follicular, medullary, or papillary thyroid cancer, non-small cell lung cancer, hepatocellular carcinoma, carcinoma of the head and neck, and renal cell carcinoma.
* To evaluate the safety of R935788 in patients with various solid tumors.
* To determine the effects of R935788 on circulating tumor cells, circulating endothelial cells and levels of phosphorylated AKT and extracellular-signal regulated kinase (ERK) in tumor samples.
* To evaluate the biochemical response to R935788 therapy in patients with thyroid malignancies and pheochromocytoma.

ELIGIBILITY

* Patients with histologically documented pheochromocytoma, follicular, medullary, or papillary thyroid cancer, colorectal cancer, non-small cell lung carcinoma (excluding squamous cell histology), hepatocellular carcinoma, carcinoma of the head and neck, as well as renal cell carcinoma) whose disease has progressed after any therapy or who have no acceptable standard treatment options.
* Radiation or chemotherapy is not permitted within 4 weeks prior to study enrollment.
* Patients must have recovered from toxicities of prior therapies to at least eligibility levels.

STUDY DESIGN

-This is an open-label, Phase II study of R935788. Patients will receive R935788 orally twice a day in 28-day cycles without interruption. Imaging studies will be obtained every 2 cycles. Following a limited dose escalation portion in each stratum, a two stage design will be used, the initial stage of which will consist of 15 to 21 patients depending on tumor type in each of 7 strata.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 3.1.1 Subjects must have histologically documented solid tumors: pheochromocytoma, follicular or papillary thyroid, colorectal, non-small cell lung (excluding squamous cell histology), hepatocellular, head and neck or renal cell origin, whose disease has progressed after any number of prior therapies or who have no acceptable standard treatment options.
* Patients with follicular or papillary thyroid cancer will be eligible if they have metastatic or unresectable, locally advanced disease which is refractory to, or not suitable for, I therapy.
* Diagnosis of malignancy must be confirmed by the Laboratory of Pathology at the Clinical Center, National Institutes of Health (NIH), prior to patient enrollment.
* 3.1.2 Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
* 3.1.3 Life expectancy of greater than 3 months.
* 3.1.4 Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* 3.1.5 Subjects must have normal organ and marrow function as defined below:
* absolute neutrophil count greater than or equal to 1,500/mcL
* platelets greater than or equal to 100,000/mcL
* total bilirubin within less than or equal to 1.5 institutional upper limit of normal (ULN)
* aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase(SGOT),alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 times ULN
* creatinine < 1.5 times ULN

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels greater than or equal to 1.5 times institutional upper limit of normal.
* 3.1.6 The effects of R935788 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for 1 month after discontinuation of the study. Women of child bearing potential must have a negative pregnancy test in order to be eligible. Should a participant or a participant's partner become pregnant or suspect she is pregnant while participating in this study, the participant should inform the Research Team immediately.
* 3.1.7 Ability to understand and the willingness to sign a written informed consent document.
* 3.1.8 Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of R935788 in patients < 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase I trials.
* 3.1.9 Patients with diagnosis of hypertension should have their blood pressure adequately controlled by medical therapy (adequate control of hypertension for the purposes of this trial is defined as systolic blood pressure < 150 mmHg or diastolic pressure < 90 mmHg).
* 3.1.10 Patients with head and neck cancer who are unable to swallow and who are gastrostomy tube (G-tube) dependent will have the tablets dissolved in water or orange juice followed by a free water or orange juice flush.

EXCLUSION CRITERIA:

* 3.2.1 Subjects who have had chemotherapy, biotherapy, or radiotherapy within 4 weeks prior to entering the study, or those who have not recovered from adverse events due to prior therapy.
* A time period of greater than or equal to 2 weeks must have elapsed since a patient was administered any investigational agent as part of a Phase 0 study (also referred to as an early Phase I study or pre-Phase I study where a sub-therapeutic dose of drug is administered) at the principal investigator's (PI's) discretion, and patients should have recovered from any toxicity from prior therapy to eligibility levels.
* 3.2.2 Patients must not have other current malignancies, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast.
* Patients who have undergone primary therapy for a prior diagnosis of cancer and are disease free for at least 3 years prior to study entry will be included in the trial.
* 3.2.3 Patients may not be receiving any other investigational agents.
* 3.2.4 Subjects with known brain metastases are excluded with the exception of those whose brain metastatic disease status has remained stable for at least 3 months since treatment of the brain metastases without steroids (except for maintenance replacement doses) or antiseizure medications.
* Patients cannot be taking enzyme-inducing anti-seizure medications (e.g., phenytoin, carbamazepine, phenobarbital, primidone, oxcarbamazepine); other seizure medications that are not considered enzyme-inducing would be permissible.
* 3.2.5 Because there is an unknown but potential risk for adverse events in nursing infants secondary to exposure to this agent, women who are breast feeding are ineligible for this study.
* 3.2.6 Patients receiving medications known to induce/inhibit cytochrome P450 3A4 (CYP3A4) will be excluded from this study.
* Patients who must initiate treatment with a CYP3A4 inhibitor while receiving R935788 will be carefully monitored.
* Inhibitors of CYP3A4 include but are not limited to:
* amiodarone,
* clarithromycin,
* erythromycin,
* imatinib,
* troleandomycin,
* ritonavir,
* indinavir,
* fluconazole,
* itraconazole,
* and ketoconazole.
* Patients should also avoid grapefruit and grapefruit juice during participation in the study.
* Patients will also be required to keep a study diary to record any side effects that occur during the study and any other medications taken.
* 3.2.7 Subjects with clinically significant illnesses which would compromise participation in the study, including, but not limited to: unstable or serious medical conditions (ongoing or active infection, symptomatic congestive heart failure [AHA Class II or worse], unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements) are excluded due to the possibility that the underlying condition may obscure the attribution of effect and adverse events with respect to the study medication and may limit study compliance.
* 3.2.8 Patients with hepatocellular cancer (HCC) may have underlying chronic infectious hepatitis as long as there is no evidence of hepatic failure and they meet the eligibility criteria.
* 3.2.9 Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with R935788.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lenders JW, Pacak K, Walther MM, Linehan WM, Mannelli M, Friberg P, Keiser HR, Goldstein DS, Eisenhofer G. Biochemical diagnosis of pheochromocytoma: which test is best? JAMA. 2002 Mar 20;287(11):1427-34. doi: 10.1001/jama.287.11.1427. PMID 11903030
- [Background] Pacak K, Eisenhofer G, Carrasquillo JA, Chen CC, Li ST, Goldstein DS. 6-[18F]fluorodopamine positron emission tomographic (PET) scanning for diagnostic localization of pheochromocytoma. Hypertension. 2001 Jul;38(1):6-8. doi: 10.1161/01.hyp.38.1.6. PMID 11463751
- [Background] Gimenez-Roqueplo AP, Favier J, Rustin P, Rieubland C, Crespin M, Nau V, Khau Van Kien P, Corvol P, Plouin PF, Jeunemaitre X; COMETE Network. Mutations in the SDHB gene are associated with extra-adrenal and/or malignant phaeochromocytomas. Cancer Res. 2003 Sep 1;63(17):5615-21. PMID 14500403
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0138.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Multi-kinase Inhibitor Fosamatinib Disodium: 200 mg BID was the administered dose for the initial part of the study and then a phase I dose escalation was added with 100 mg as the starting dose.
Period: Overall Study
Arm/Group | Multi-kinase Inhibitor Fosamatinib Disodium
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multi-kinase Inhibitor Fosamatinib Disodium
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.73 (9.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response is assessed by the RECIST (response criteria in solid tumors)criteria. A complete response (CR) is disappearance of all target lesions , partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions, and stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 24 months
Measure: Number; unit: Participants
Arm/Group | Multi-kinase Inhibitor Fosamatinib Disodium
Number analyzed (Participants) | 37
Participants
  Complete response | 0
  Partial Response | 0
  Progressive disease | 26
  Stable disease | 11

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 23 months
Measure: Number; unit: Participants
Arm/Group | Multi-kinase Inhibitor Fosamatinib Disodium
Number analyzed (Participants) | 37
Participants | 37

ADVERSE EVENTS:
Arm/Group | Multi-kinase Inhibitor Fosamatinib Disodium
Serious Adverse Events (participants affected / at risk) | 11/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-kinase Inhibitor Fosamatinib Disodium (N=37)
Alkaline phosphatase (Investigations) | 1 (1)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 1 (1)
Death not associated with CTCAE term::Death NOS (General disorders) | 2 (2)
Death not associated with CTCAE term: Death Progression NOS (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pharynx (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway (Infections and infestations) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Pain::Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-kinase Inhibitor Fosamatinib Disodium (N=37)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 22 (57)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 23 (66)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 29 (77)
Alkaline phosphatase (Investigations) | 17 (32)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bicarbonate, serum low (Metabolism and nutrition disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Investigations) | 13 (29)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
CPK (creatine phosphokinase) (Investigations) | 7 (15)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 10 (19)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5 (7)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Creatinine (Investigations) | 4 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Dermatology/Skin - Other (Specify, laceration) (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (11)
Dizziness (Nervous system disorders) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Edema::head and neck (General disorders) | 1 (1)
Edema limb (General disorders) | 1 (1)
Extremity-lower (gait/walking) (General disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (12)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (4)
Glucose, serum-low (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Investigations) | 24 (47)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory::Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 11 (19)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Renal and urinary disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Eye NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Neck NOS (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 3 (3)
Infection with unknown ANC::Sinus (Infections and infestations) | 1 (1)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Leukocytes (total WBC) (Investigations) | 15 (37)
Lymphopenia (Investigations) | 25 (62)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 16 (29)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 (8)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8)
Neuropathy - motor (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4 (6)
Pain::Other (Specify, pain-epigastric) (General disorders) | 1 (1)
Paib:: Abdomen NOS (General disorders) | 4 (5)
Pain::Abdomen NOS (Gastrointestinal disorders) | 1 (1)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Eye (Eye disorders) | 1 (2)
Pain::Head/headache (Nervous system disorders) | 4 (4)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 10 (16)
Platelets (Investigations) | 6 (8)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 6 (8)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6 (6)
Proteinuria (Renal and urinary disorders) | 1 (2)
Rigors/chills (General disorders) | 4 (5)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 20 (33)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 3 (5)
Vision-blurred vision (Eye disorders) | 1 (1)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Weight loss (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No